CLINICAL TRIAL: NCT03236714
Title: Awareness and Compliance Among Health Professionals of the Preoperative
Brief Title: Awareness and Compliance Among Health Professionals of the Preoperative Fasting Period
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assist.Prof, Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-005
Record Dates: First submitted 2017-07-24; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Preoperative Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative fasting is mandatory for anesthetic induction. This period of fasting is probably greater due to delays in the surgical theater and changes in daily operation schedules.Investigators want to resarch between the prescribed and the actual preoperative fasting time.

DETAILED DESCRIPTION:
Before surgery, the patients will be asked to liquid, solid fasting times.and whether information is given about the fasting period.In addition, the appropriateness of health personnel to new guidelines for preoperative fasting will be evaluated.At the end of the study, the desired duration of fasting, clinical practice and trends of health personnel will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 day and 80 years
* Elective surgery
* Oral fed
* American Society of Anesthesiologists score of 1 or 3

Exclusion Criteria:

* Intensive care patient
* Parenteral nutrition
* Emergency surgery

Ages: 1 Day to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients planning elective surgery according to the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-05 (Estimated)

PRIMARY OUTCOMES:
The patients' preoperative fasting period | one time in two months
  Determination of fasting period before surgery trends of new guidelines for preoperative fasting.
Training of health workers | one time in two months
  Determining health personnel's application

CONTACTS AND LOCATIONS:
Locations (1):
- Hakan Tapar, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No